CLINICAL TRIAL: NCT05428787
Title: Resynchronization in Patients With Ambulatory Heart Failure in Atrial Fibrillation Trial Undergoing Pace and Atrioventricular Node Ablation Strategy With Left Bundle Branch Area Pacing Compared With Biventricular Pacing
Brief Title: Resynchronization in Patients With HF in AF Trial Undergoing Pace & AVNA Strategy With LBBAP Compared With BiV Pacing
Acronym: RAFT-P&A
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Habib Khan (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Habib Khan, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3819
Record Dates: First submitted 2022-05-10; First posted 2022-06-23 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Heart Failure; Cardiomyopathies
Keywords: LBBAP; Conductions system pacing; atrial fibrillation; pace and ablate; AV node ablation; CRT; BiV-CRT
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Resynchronization Therapy + AV node ablation (Active Comparator): The active comparator group will be treated with CRT followed by an Atrioventricular Node Ablation.
  Interventions: Procedure: CRT; Procedure: AV node ablation
- Left Bundle Branch Area Pacing + AV node ablation (Experimental): The experimental group will be treated with LBBAP followed by an Atrioventricular Node Ablation.
  Interventions: Procedure: Left Bundle Branch Area Pacing; Procedure: AV node ablation

INTERVENTIONS:
Procedure: Left Bundle Branch Area Pacing — The patients will be allocated by randomization to receive the intervention of Left Bundle Branch Area Pacing
  Other Names: LBBAP
  Arms: Left Bundle Branch Area Pacing + AV node ablation
Procedure: CRT — The patients will be allocated by randomization to receive the intervention of CRT.
  Arms: Cardiac Resynchronization Therapy + AV node ablation
Procedure: AV node ablation — AV node ablation after 4 weeks of CRT implant or LBBAP implant.

SUMMARY:
This trial will compare two management strategies for HF patients with Atrial Fibrillation. The active control group will undergo BiV pacing, followed by an AV node ablation. The experimental group will undergo LBBAP, followed by an AV node ablation.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind, control trial with follow up visits at 6- and 12-months following randomization. Patients will be randomized in a 1:1 allocation to either the control group [optimal medical therapy (OMT) + CRT + ANVA] or the treatment group [OMT + LBBAP + ANVA]. Randomization will be stratified by site and LVEF. In each group, the patient will undergo the pacing procedure (CRT or LBBAP) within 10 working days of randomization. They will be assessed by a physician one week after the CRT procedure, and if eligible, they will undergo an AVNA within 1-4 weeks. Success of these treatment plans will be evaluated primarily based on the change in NT-proBNP from baseline to 6- and 12-month follow ups. At baseline and follow up visits study staff and physicians will collect participants' medical history, complete a Physical Exam and an NYHA Class Assessment, a medication assessment, and a 6 Minute Walk Test. Participants will also be asked to complete Quality of Life Questionnaires (Minnesota Living with Heart Failure Questionnaire (MLHFQ) score, KCCQ and EQ-5D-5L), have an ECG and TTE performed if they have not had one performed recently, non- invasive hemodynamic measurements (if available), and complete routine bloodwork and an NT-proBNP test. The adequacy of HF treatment will be assessed clinically, and medications optimized and recorded. Device diagnostics will be assessed and recorded as to whether there are arrhythmias and to determine the appropriateness of device programming. Secondary study outcomes include QoL scores (MLHFQ, KCCQ and EQ-5D), as well as 6MWT distance, and change in echocardiogram parameters (including change in LVESV index from baseline, change in global longitudinal LV systolic strain from baseline, and change in LVEF from baseline at 6-month and 12-month followup). Secondary outcomes also include radiation exposure between LBBAP and CRT, feasibility of achieving conduction system pacing with LBBAP compared to CRT, and acute and long-term hemodynamic change due to either CRT or LBBAP (i.e., non-invasive hemodynamic measurements before and after AV node ablation including systolic BP, diastolic BP, cardiac output, stroke volume, total peripheral resistance, and pulse pressure).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atrial fibrillation (AF) where AVNA is being considered with or without a pacemaker

   1. Are on optimal heart failure therapies for ≥4 weeks
   2. NYHA class I-IVa
2. Patients deemed not appropriate for rhythm control strategy (only for rate control strategy).

   1. Failed Ablation (≥1 failed ablation attempt)
   2. Refractory or intolerant to Antiarrhythmic drugs AADs or rate control medications
   3. Patient choice not to have rhythm control strategies
   4. Being considered for AVNA
3. Patients with baseline NT-proBNP>600 or >400 if HF hospitalization within 12 months.

Exclusion Criteria:

1. In-hospital patients with acute cardiac or non-cardiac illness that requires intensive care
2. Acute coronary syndrome (including MI) or Coronary revascularization (CABG or PCI) <3 months
3. Uncorrected or uncorrectable primary moderate to severe valvular disease
4. TAVI < 3 months
5. Restrictive, or reversible form of cardiomyopathy, cardiac amyloidosis
6. Severe primary pulmonary disease such as cor pulmonale, irreversible lung disease requiring inhalers, oxygen supplementation
7. Pulmonary hypertension (Mean pulmonary pressure is ≥35 mm Hg)
8. Patients with a life expectancy of less than one year from non-cardiac cause
9. Patients included in other clinical trials that will affect the objectives of this study or have competing interests
10. Those unable or unwilling to provide informed consent unless supported by legal power of attorney
11. Active malignancy with likelihood of survival <1 year
12. NYHA class IVb

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in NT-proBNP from baseline to 6-month follow-up | baseline and 6 months
  Comparison between NT-proBNP measurement at baseline and 6-month follow-up

SECONDARY OUTCOMES:
Event rates of the composite outcome of heart failure events and all-cause mortality | 12 months
  HF and mortality data will be collected throughout the duration of the study
Change in QoL - MLHFQ | baseline, 6 months and 12 months
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) score is used to measure quality of life. The MLHFQ consists of 21 questions answered on a 0-5 likert scale, with higher scores indicating a stronger impact of heart failure on QoL.
Change in QoL - KCCQ | baseline, 6 months and 12 months
  Cardiomyopathy Questionnaire (Kansas City) (KCCQ-12) measures how heart failure impacts a patient's quality of life. The questionnaire measures frequency and burden of heart failure symptoms as well as physical and social limitations related to heart failure using a likert scale of 0-100, with higher scores indicating better health.
Change in QoL - EQ-5D | baseline, 6 months and 12 months
  EuroQol- 5 Dimension measures health related quality of life using a Level 1-5 component scale. A lower score indicates better health related quality of life. The EQ-5D also contains the EQ VAS, a 0-100 self reported scale where 100 indicates best health imaginable.
Change 6MWT distance | baseline, 6 months and 12 months
  Change in distance walked in the 6MWT from baseline to 6-month and 12-month follow-up
Change in echocardiogram parameters - Left Ventricular End Systolic Volume index (LVESVi) | baseline, 6 months and 12 months
  Compared from baseline to 6-month and 12-month follow-up. A lower LVESVi indicates a trend towards normal volumes and a higher LVESVi indicates ventricle dilation compared to the normal population.
Change in echocardiogram parameters - Left Ventricle (LV) Global Longitudinal strain | baseline, 6 months and 12 months
  Compared from baseline to 6-month and 12-month follow-up. A lower LV Global Longitudinal strain indicates stronger left ventricular contraction.
Change in echocardiogram parameters - Left Ventricular Ejection Fraction (LVEF) | baseline, 6 months and 12 months
  Compared from baseline to 6-month and 12-month follow-up. An increase in LVEF indicates stronger function of the left ventricle.
Radiation exposure at device implant | During Surgical Intervention
  Exposure time collected at device implant visits

CONTACTS AND LOCATIONS:
Overall Officials: Habib Khan, MBBS, PhD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No